CLINICAL TRIAL: NCT03791125
Title: Randomized, Double-blind, Placebo-controlled, Single-dose Escalation, Evaluation of Safety, Tolerability, and Pharmacokinetic Properties of Salvianolic Acid A Tablets in Healthy Volunteers
Brief Title: Phase I Single-dose Escalation Clinical Trial of Salvianolic Acid A Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Shandong Huizhi Pharmaceutical Technology Co., Ltd. (Unknown); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Cui Yimin, Director of Pharmacy, M.D. and Ph.D., Peking University First Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018028
Record Dates: First submitted 2018-11-15; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Neuropathy of Diabetes
MeSH Terms: interventions — salvianolic acid A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: Salvianolic Acid A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Salvianolic Acid A — 4 anticipated doses are 30 mg, 90 mg, 180 mg and 270 mg, respectively. All of these are single-dose study.
  Arms: Experimental
Drug: Placebo Oral Tablet — Placebo tablets containing no salvianolic acid A will be given to healthy subjects.
  Arms: Placebo

SUMMARY:
Salvianolic acid A has a variety of pharmacological effects, such as: anti-oxidation, scavenging oxygen free radicals, anti-fibrosis, anti-myocardial ischemia, anti-coagulation, anti-thrombosis, anti-tumor, etc. Professor Du Guanhua, at Institue of Materia Medica, Chinese Academy of Medical Sciences, first discovered that salvianolic acid A can alleviate diabetic complications and improve patients' quality of life. With the support of major national science and technology projects, the preclinical research work of salvianolic acid A was completed, and the application was approved by the State Food and Drug Administration (Clinical Approval No.: 2016L06293). Peking University First Hospital was used as the research unit. This study is the first human clinical trial of the drug. The project leader of this study is Professor Cui Yimin from Peking University First Hospital. The sponsor of this project is Shandong Huizhi Pharmaceutical Technology Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

* 1) Gender: male or female, healthy volunteers; 2) Age: 18~45 years old; 3) Weight: Male subjects need to weigh ≥ 50kg, female subjects should have ≥ 45kg, body mass index [BMI = weight (kg) / height 2 (m2)] in the range of 19 ~ 25 kg / m2; 4) Subjects must give informed consent to the trial prior to the trial and voluntarily sign a written informed consent form; 5) The subject is able to communicate well with the investigator and is able to complete the trial in accordance with the protocol.

Exclusion Criteria:

* (1) Hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus and syphilis positive; (2) alcoholics; (3) subjects who took any drug or long-term use of drugs within 2 weeks before screening (4) Blood donors within 3 months prior to the trial; (5) participated in any drug clinical trial within 3 months prior to screening; (6) had a clear history of allergic disease; (7) had central nervous system, cardiovascular Systematic, kidney, liver, digestive tract, lung disease, metabolic and skeletal muscle system with a clear history or other significant disease; (8) pregnant, lactating women; (9) other factors not suitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events | 7 days
Percentage of participants with change from baseline in vital signs | 7 days
  Heart rate, Blood Pressure，auxillary temperature
Change from baseline in electrocardiograms (ECGs) | 7 days
  PR interval, QT interval, QTc interval, QTcF, and rhythm abnormalities
Percentage of participants with change from baseline in clinical laboratory parameters | 7 days
  blood routine, urine routine, biochemical parameters of blood and urine，coagulation tests
PK profile of Salvianolic acid A following administration of multiple doses assessed by area under the curve [AUC] | 2 days
PK profile of Salvianolic acid A following administration of multiple doses assessed by maximum observed concentration [Cmax] | 2 days
PK profile of Salvianolic acid A following administration of multiple doses assessed by time of occurrence of Cmax [tmax] | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy, Base for Clinical Trial, Peking University First Hospital, Beijing, Beijing Municipality, China